CLINICAL TRIAL: NCT04383834
Title: 2017-1538: A 3-years Investigator Initiated Study to Evaluate the Soft Tissue Health and Stability in the Mandible and/or Maxilla Using the NobelActive® TiUltra™ and On1™ Base/Xeal™
Brief Title: A 3-YEAR CLINICAL INVESTIGATION ON THE NOBEL ACTIVE® TIULTRA™ IMPLANT AND ON1™ BASE XEAL1™ _____________________________________________________________
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Giacomo Fabbri (Network)
Responsible Party: Sponsor-Investigator, Giacomo Fabbri, Giacomo Fabbri, Studio Ban Mancini Fabbri
Organization: Studio Ban Mancini Fabbri (Network)
Other Study IDs: 2017-1538
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: to Study Soft Tissue Health and Stability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 47 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: NobelActive® TiUltra™ implants and On1™ Base/Xeal™ along with On1 components — The NobelActive® TiUltra™ implant is an ultra-hydrophilic multi-zone anodized implant surface. NobelActive® TiUltra™ features a gradual change in topography, from a minimally rough non-porous nanostructured implant collar to a moderately rough porous apex: more than roughness. NobelActive® TiUltra™ collar features surface chemistry and topography that promote early osseointegration and are designed to support bone stability. In addition, the Protective Layer preserves the pristine surface chemistry and hydrophilicity.
  The second new product is the Base/Xeal™ new surface, which is covered by a titanium oxide layer, created by electrochemical anodization of a titanium machined component, resulting in a yellow hue nano-structured surface.

SUMMARY:
Soft tissue thickness, using IOS, between implant insertion (baseline) and 3-year follow-up has no changes

ELIGIBILITY:
Inclusion Criteria:

.The subject inclusion criteria are listed below. The subject is at least 18 years of age (or age of consent) and has passed cessation of growth.

Obtained informed consent from the subject. The patient is willing and able to comply with all study related procedures (such as exercising oral hygiene and attending all follow-up procedures).

The subject shall be healthy and compliant with good oral hygiene. Full-mouth bleeding score (FMBS) lower than 25 %[10]. Full-mouth plaque score (FMPI) lower than 20% [11]. Suitable for implant treatment in the posterior, pre-molar area in the mandible or maxilla.

The subject shall have a favorable and stable occlusal relationship. In need of one single tooth replacement Healed sites in need for implant placement (i.e. minimum of 6 weeks post extraction).

The implant sites are free from infection and extraction remnants. The subject is suitable for a 1-stage surgical procedure. Sufficient amount of buccal and lingual keratinized mucosa. The healed sites eligible will have natural teeth as neighboring structures. The subject is in such a physical and mental condition that a 3-year follow up period can be carried out without foreseeable problems.

The subject has a sufficient amount of bone for placing NobelActive TiUltra with a length of at least 7 mm.

The following subject inclusion criteria apply at time of surgery:

Primary implant stability as assessed by manual hand testing.

Exclusion Criteria:

* The subject is not able to give her/his informed consent of participating. Health conditions, which do not permit the surgical (including anesthesia) or restorative procedure.

Reason to believe that the treatment might have a negative effect on the subject's overall situation (psychiatric problems), as noted in subject records or in subject history.

Any disorders in the planned implant area such as previous tumors, chronic bone disease or previous irradiation in the head/neck area.

Infections in the planned implantation site or adjacent tissue. Acute, untreated periodontitis in the planned implantation site or adjacent tissue.

Any ongoing application of interfering medication (steroid therapy, bisphosphonate, etc.).

Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake or A1c level above 8%.

Alcohol or drug abuse as noted in subject records or in subject history. Smoking less 10 cigarettes/day. Fresh extraction sites (up to 6 weeks). Severe bruxism or other destructive habits. Pregnant or lactating women at the time of implant insertion. Previous bone augmentation (lateral and/or vertical). Soft tissue augmentation less than 2 months before implant placement. Subject has allergic or adverse reactions to the restorative material

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects, at least 18 years old, in need of one single restoration in the posterior region of the maxilla and/or the mandible.
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
A 3-years Investigator initiated study to evaluate the soft tissue health and stability in the mandible and/or maxilla using the NobelActive® TiUltra™ and On1™ Base/Xeal™ | 47 months (8 months enrolment + 36 months follow up + 3 months study closure)
  Soft tissue thickness, using IOS, between implant insertion (baseline) and 3-year follow-up has no changes

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Fabbri, Dentist, Principal Investigator — Studio Ban Mancini Fabbri
Locations (1):
- Studio Ban Mancini Fabbri, Cattolica, Rimini, Italy

IPD SHARING:
Plan to Share IPD: No